CLINICAL TRIAL: NCT05248217
Title: Assessment of Burnout Syndrome and Smartphone Addiction in Healthcare Workers Actively Working During the COVID-19 Pandemic
Brief Title: Burnout, Covid 19, Smarthphone Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: burnout smarthphone1
Record Dates: First submitted 2022-02-18; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Burn Out; Addiction, Smartphone
Keywords: burnout; covid-19; healthcare workers; smarthphone addiction
MeSH Terms: conditions — Burnout, Psychological; Internet Addiction Disorder; COVID-19 | interventions — Health Personnel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthcare workers (Other): doctors, nurses, medical secretaries, security guards, and cleaning staff
  Interventions: Behavioral: healthcare workers

INTERVENTIONS:
Behavioral: healthcare workers — healthcare

SUMMARY:
We investigate burnout syndrome and smartphone addiction in healthcare workers, including doctors, nurses, medical secretaries, security guards, and cleaning staff, who have been actively working from the beginning of the COVID-19 pandemic. target population included 1190 healthcare workers, from which a total of 183 agreed to participate in the study and met the inclusion criteria for participation. A sociodemographic data form, the Maslach Burnout Inventory, and the Smartphone Addiction Scale-Short Version were used as the data collection tools.

DETAILED DESCRIPTION:
Significant differences in burnout syndrome were found in doctors and nurses. A relationship was observed between emotional burnout (EB), desensitization, and smartphone addiction, as well as between doctor and nurse group, and smartphone addiction. According to the linear regression analysis, it was determined that 17% of the change in the smartphone addiction score was related to age and 16% to master education level.Doctors and nurses experience the highest rate of burnout syndrome and smartphone addiction, and EB and desensitization were more likely to have smartphone addiction. Age and high education can affect smarthphone addiction

ELIGIBILITY:
Inclusion Criteria:

1. Being older than 18 years of age
2. Working as medical staff
3. Having no systemic or psychiatric disorders
4. No psychotropic substances use
5. No alcohol or substance use

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
maslach burnout scale | 30 minutes
  This tool was developed by Maslach and Jackson (1981), and the validity and reliability study of its Turkish version was conducted by Ergin (1992). The inventory has 22 items, which are scored on a 5-point Likert-type scale with anchors of 0 (never) and 4 (always). The MBI has three subscales: emotional burnout (9 items), desensitization (5 items), and low personal success (8 items

SECONDARY OUTCOMES:
smarthphone addiction scale | 15 minutes
  This 6-point Likert-type scale was developed by Kwon et al. to assess the risk of smartphone addiction. Total scale scores range from 10 to 60, with higher scores indicating higher risk of addiction. This is a single factor scale, and it has no subscales. The Cronbach's alpha coefficient of internal consistency and concurrent validity was 0.91 for the original scale

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdogan University, Rize, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No